CLINICAL TRIAL: NCT05519852
Title: Quality of Life Response to Pilates Physical Activity in Sickle Cell Disease
Brief Title: Pilates Physical Activity in Sickle Cell Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003820
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): this pilates group (20 patients) will be trained 30 minutes of pilates (before it there will be warm up period and after it there will be cooldown period , each will be 5 minutes). the pilates will be repeated five sessions per the week for 3 months
  Interventions: Behavioral: Pilates training
- control group (No Intervention): The patients will not receive training (20 patients)

INTERVENTIONS:
Behavioral: Pilates training — the pilates group (20 patients) will be trained 30 minutes of pilates exercise (before it there will be warm up period and after it there will be cooldown period , each will be 5 minutes). the pilates will be repeated five sessions per the week for 3 months
  Arms: Pilates group

SUMMARY:
Sickle cell anemia (SCA) is a life-threatening hereditary hemoglobinopathy characterized by hemoglobin (Hb) polymerization that affects many people worldwide.Reduced physical capacity is common in people with SCA. Pilates is a form of physical activity that recently used in clinicial practice

DETAILED DESCRIPTION:
SCA patients (40 patients) with ages more than 18 years will join randomly the pilates group (20 patients) or control non exercised group (20 patients). Pilates will be trained 30 minutes (before it there will be warm up period and after it there will be cooldown period , each will be 5 minutes). the pilates will be repeated five sessions per the week for 3 months

ELIGIBILITY:
Inclusion Criteria:

* sedentary sickle disease patients from both both sexes in medical stable condition

Exclusion Criteria:

* cardiac complaints, pregnant women, patients who smoke or drink alchols

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | It will be measured after 12 weeks
  it assess sleep quality

SECONDARY OUTCOMES:
six minutes walking distance | It will be measured after 12 weeks
  it will assess physical capacity
quadriceps strength | It will be measured after 12 weeks
  it will assess the muscular strength of dominant quadriceps
hand grip strength | It will be measured after 12 weeks
  it will assess the muscular strength of dominant hand grip
physical component summary of short-form-36 questionnaire | It will be measured after 12 weeks
  it will assess physical health
mental component summary of short-form-36 questionnaire | It will be measured after 12 weeks
  it will assess mental health
beck depression inventory | It will be measured after 12 weeks
  it is a questionnaire assessing depression

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, Principal Investigator — Lecturer, Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt